CLINICAL TRIAL: NCT02510443
Title: Survey on Use and Characteristics of Definitive Contraception With ESsure®
Brief Title: Observational Study on Contraception With Essure in France
Acronym: SUCCES II
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Hôpital André Mignot Centre Hospitalier de Versailles (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18097; ES0810FR (Other: Company Internal)
Record Dates: First submitted 2015-06-15; First posted 2015-07-29 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: Permanent contraception method; Contraceptive device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BAY1454032: All subjects who give their consent and meet the eligibility criteria will be scheduled for an insert placement procedure
  Interventions: Device: ESS305 (Essure, BAY1454032)

INTERVENTIONS:
Device: ESS305 (Essure, BAY1454032) — Bilateral insert placement

SUMMARY:
Using a very broad survey, the objective is to confirm the effectiveness of the Essure method, and to obtain more information on the conditions of use as well as on the methods used during the 3-month check-up, as well as the 12-month, 24-month and 5-year follow-up on patients.

DETAILED DESCRIPTION:
The study is a prospective epidemiological survey to collect local real life data on patients under routine pratice

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years old,
* Scheduled for Essure procedure
* Patient who has been given appropriate information about the study objectives and procedures and who has given her consent.

Exclusion Criteria:

* Patients with contraindications as listed in the current Instruction For Use (IFU) will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients concerned are adult women wishing to undergo tubal sterilization for contraceptive purposes, in accordance with legal provisions, who had given their consent for collection of the data.
Sampling Method: Non-Probability Sample
Enrollment: 2644 (Actual)
Dates: Start 2008-06-23 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Number of patients being satisfied with successful Essure procedure having no complications at 5 years | At 5 years
  Patient satisfaction will be assessed on a Likert scale. Complications are migration/expulsion of Essure, infection. Pregnancy will be measured at any time Point.

SECONDARY OUTCOMES:
Number of patients with moderate or important pain when placement is performed | At initial visit
  Visual Analogue Scale (VAS) use to report the pain from 0 (no pain) to 10 (maximal pain). Moderate pain will range from 4 to 6 and important pain will range from 7 to 10 on the VAS.
Number of unsatisfied patients | Up to 5 years
Number of satisfied patients at 3, 12 and 24 months | At 3 ,12 and 24 months
  Patients satisfaction assessed by Likert scale.
Number of examinations by patients | At 3 months
Number of good insert position by implant and patients with success in final result of the procedure | At 3 months
Causes of unsatisfied patients | Up to 5 years
  Possible causes of unsatisfaction : pregnancy, regret of the patient,migration/expulsion of Essure,or infection
Type of examinations by patients | At 3 months
  Ultrasound transvaginale, radiography, or hysterosalpingography (HSG)
Number of patients with regrets | At 12 months, 24 months and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Le Chesnay, France